CLINICAL TRIAL: NCT04633629
Title: Interest of Lung Ultrasound (LUS) in Therapeutic Adaptation of Patients Hospitalized in Medical Department for Acute Heart Failure (AHF).
Brief Title: LUS in Acute Heart Failure Therapeutic Adaptation
Acronym: EPPICA
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC20.328; 2020-A02413-36 (Other: ID RCB)
Record Dates: First submitted 2020-09-08; First posted 2020-11-18 (Actual); Last update posted 2020-11-18 (Actual); Status verified 2020-11

CONDITIONS: Acute Heart Failure; Pulmonary Congestion
Keywords: Lung Ultrasound; Diuretics; Medical department

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with acute heart failure: Patients hospitalized for acute heart failure in medical department.
  Interventions: Other: Lung ultrasound

INTERVENTIONS:
Other: Lung ultrasound — We will perform daily a lung ultrasound to evaluate pulmonary congestion by counting B-lines.

SUMMARY:
Evaluate lung ultrasound aspect according to diuretics dosage evolution in patients hospitalized for acute heart failure.

DETAILED DESCRIPTION:
EPPICA is an observational and prospective cohort study. The study goal is to evaluate LUS aspect evolution according to diuretics dosage in patients hospitalized for acute heart failure.

ELIGIBILITY:
Inclusion Criteria:

* Acute heart failure diagnosed by a senior physician in the medical department, with a confirmation of a second senior physician.
* Hospitalised in the medical department.
* No objection from the patient of his trusted person.

Exclusion Criteria:

* Administrative supervision or deprived of their liberty
* Pulmonary conditions distracting lung ultrasound (pneumonectomy, pulmonary fibrosis)
* Chronically dialysed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged over 18, hospitalized from the emergency department in the medical department for acute heart failure.
Sampling Method: Non-Probability Sample
Enrollment: 94 (Estimated)
Dates: Start 2020-12 (Estimated); Primary Completion 2021-05 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Lung ultrasound aspect according to diuretics dosage evolution. | LUS will be performed daily during the whole hospitalisation length (on average 7 days).
  B-lines number on LUS

SECONDARY OUTCOMES:
Lung ultrasound aspect according to clinical signs of acute heart failure (crackling auscultation or lower limbs edema) | LUS and clinical examination will be performed daily during the whole hospitalisation length (on average 7 days).
  B-lines number on LUS
Lung ultrasound aspect according to acute kidney injury (based on plasmatic creatinine levels). | LUS will be performed daily during the whole hospitalisation length (on average 7 days). Plasmatic creatinine measure will be performed at least weekly.
  B-lines number on LUS
Lung ultrasound aspect according to early prognosis (re-hospitalisation or mortality within 30 days after discharge) | LUS will be performed daily during the whole hospitalisation length (on average 7 days). Patient will be called 30 days after discharge.
  B-lines number on LUS
Feasibility of daily LUS in medical department. | LUS will be performed daily during the whole hospitalisation length (on average 7 days).
  Number of LUS performed compared to number of hospitalisation days.
Interest of LUS compared to clinical examination at discharge. | LUS and clinical examination will be performed daily during the whole hospitalisation length (on average 7 days).
  B-lines at discharge compared to clinical signs of acute heart failure.

CONTACTS AND LOCATIONS:
Overall Officials: Perrine Dumanoir, Doctor, Principal Investigator — University Hospital, Grenoble

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ohman J, Harjola VP, Karjalainen P, Lassus J. Focused echocardiography and lung ultrasound protocol for guiding treatment in acute heart failure. ESC Heart Fail. 2018 Feb;5(1):120-128. doi: 10.1002/ehf2.12208. Epub 2017 Sep 28. PMID 28960894
- [Background] Coiro S, Rossignol P, Ambrosio G, Carluccio E, Alunni G, Murrone A, Tritto I, Zannad F, Girerd N. Prognostic value of residual pulmonary congestion at discharge assessed by lung ultrasound imaging in heart failure. Eur J Heart Fail. 2015 Nov;17(11):1172-81. doi: 10.1002/ejhf.344. Epub 2015 Sep 29. PMID 26417699
- [Background] Gargani L, Pang PS, Frassi F, Miglioranza MH, Dini FL, Landi P, Picano E. Persistent pulmonary congestion before discharge predicts rehospitalization in heart failure: a lung ultrasound study. Cardiovasc Ultrasound. 2015 Sep 4;13:40. doi: 10.1186/s12947-015-0033-4. PMID 26337295
- [Background] Platz E, Merz AA, Jhund PS, Vazir A, Campbell R, McMurray JJ. Dynamic changes and prognostic value of pulmonary congestion by lung ultrasound in acute and chronic heart failure: a systematic review. Eur J Heart Fail. 2017 Sep;19(9):1154-1163. doi: 10.1002/ejhf.839. Epub 2017 May 30. PMID 28557302
- [Background] Volpicelli G, Caramello V, Cardinale L, Mussa A, Bar F, Frascisco MF. Bedside ultrasound of the lung for the monitoring of acute decompensated heart failure. Am J Emerg Med. 2008 Jun;26(5):585-91. doi: 10.1016/j.ajem.2007.09.014. PMID 18534289
- [Background] Rusu DM, Siriopol I, Grigoras I, Blaj M, Ciumanghel AI, Siriopol D, Nistor I, Onofriescu M, Sandu G, Cobzaru B, Scripcariu DV, Diaconu O, Covic AC. Lung Ultrasound Guided Fluid Management Protocol for the Critically Ill Patient: study protocol for a multi-centre randomized controlled trial. Trials. 2019 Apr 25;20(1):236. doi: 10.1186/s13063-019-3345-0. PMID 31023358